CLINICAL TRIAL: NCT01947530
Title: Pilot Study Using Combined Virtual 4-D EM Tip-Tracked Devices and Endobronchial Ultrasound (EBUS)in the Diagnosis of Peripheral Pulmonary Nodules
Brief Title: Study Using Combined Virtual 4-D Electromagnetic (EM) Tip-Tracked Devices & EBUS in Diagnosis of Lung Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-5056-B
Record Dates: First submitted 2013-09-06; First posted 2013-09-20 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

ARMS (2):
- Navigational Bronch/Standard Bronch (Active Comparator): Patient will have first the Navigational Bronchoscopy then the standard bronchoscopy completed.
  Interventions: Procedure: Navigational Bronchoscopy; Procedure: Standard Bronchoscopy
- Standard Bronch/Navigational Bronch (Active Comparator): Patient will first have a standard bronchoscopy then a navigational bronchoscopy completed.
  Interventions: Procedure: Navigational Bronchoscopy; Procedure: Standard Bronchoscopy

INTERVENTIONS:
Procedure: Navigational Bronchoscopy
  Other Names: 4-D EM Tip-tracked Devices; Veran Navigational System
Procedure: Standard Bronchoscopy
  Other Names: Standard Bronchoscope

SUMMARY:
The purpose of this study is to determine the safety and biopsy yield of EM Tip Tracked devices compared to standard bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient aged 18 and older, able to sign an informed consent and is scheduled for flexible bronchoscopy with biopsies of peripheral nodules. Patient needs to have a recent chest CAT scan within last 4 weeks or will obtain a chest CAT scan prior to bronchoscopy.

Exclusion Criteria:

* Pulmonary nodules less than 1.0 cm
* patients must be able to tolerate general anesthesia
* patients with significant coagulopathy having International Ratio (INR)>2.0 or Prothrombin Time (PTT) >2x normal
* patients unable to tolerate bronchoscopy
* pregnant patients or patients who believe they are pregnant
* patients with implantable devices susceptible to Radio Frequency (RF) fields
* severely obese patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09; Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Observe yield of EM Tip-tracked Devices compared to standard bronchoscopy | up to 1 year
  This information will be gathered from the pathology report. This report will be completed as soon as possible after the procedure.

SECONDARY OUTCOMES:
Observe safety of EM Tip-tracked devices in the collection of samples for diagnosis of peripheral nodules | up to 1 year
Total virtual bronchoscopy time | Day 1
  Information will be gathered at time of procedure
Total procedure time | Day 1
  This information will be gathered at the time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada